CLINICAL TRIAL: NCT02125006
Title: The Effect of an Inter-Disciplinary Program, Including Mindfulness-Based Stress Reduction, on Psychosocial Function, Pain Perception, Disability and Quality of Life in Breast Cancer Survivors With Chronic Neuropathic Pain
Brief Title: The Effect of an Inter-Disciplinary Program, Including MBSR, in Breast Cancer Survivors With Chronic Neuropathic Pain
Acronym: InDepth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Breast Cancer Foundation (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20130525-01H
Record Dates: First submitted 2014-04-23; First posted 2014-04-29 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer; Painful Neuropathy; Chronic Pain; Worries; Pain or Disability; Quality of Life
Keywords: Mindfulness; Breast Cancer; Painful Neuropathy; Chronic Pain; fMRI; Disability; Quality of Life; Cytokines; Cortisol
MeSH Terms: conditions — Breast Neoplasms; Neuropathy, Painful; Chronic Pain; Pain | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interdisciplinary program including MBSR (Experimental): Participants assigned to this group will be enrolled in an Mindfulness-Based Stress Reduction (MBSR) program following medical treatment optimization. The MBSR program will be composed of eight weekly 2.5 hour sessions and one 6 hour session midway through the course.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Wait-listed Control Group (No Intervention): Participants assigned to this group after medical treatment optimization will act as wait-list controls for the MBSR group. They will be enrolled in the MBSR workshop 3 months after the corresponding intervention group completes the program.

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — Consists of eight weekly 2.5 hour sessions and one 6 hour session midway through the course. All sessions will be conducted by a psychologist or social worker with experience in chronic pain, formal MBSR training and 5 years of experience leading MBSR groups. To assess therapist adherence to the protocol, sessions will be recorded. A random selection of 50% of sessions will be rated by an MBSR trainer who completed the University of Massachusetts Centre for Mindfulness in Medicine, Health Care and Society Teacher Development Intensive using a checklist of specified treatment components. A percentage score for each session rated will be calculated to determine therapist adherence.
  Arms: Interdisciplinary program including MBSR

SUMMARY:
Chronic neuropathic pain is a common problem for breast cancer survivors. Even with the best medical treatment, some survivors continue to experience disabling pain. It is well-established that an interdisciplinary approach is key to the treatment of some types of chronic pain, but little research has been done on the effectiveness of interdisciplinary treatments for cancer survivors with chronic neuropathic pain. The investigators will evaluate the effectiveness of an interdisciplinary approach combining medical treatment and mindfulness-based stress reduction (MBSR) to reduce disability and improve quality of life among breast cancer survivors with chronic neuropathic pain. The investigators will also evaluate the impact of the program on psychological distress, pain cognitions, biomarkers of stress and immune function, cognitive function, as well as brain structure and function.

DETAILED DESCRIPTION:
The investigators will recruit 108 adult women survivors of breast cancer living with chronic neuropathic pain. All will have their medical treatment optimized by a pain medicine specialist before being randomly assigned to either an 8-week group MBSR program or a wait-list. All participants will complete self-report questionnaires, provide a hair sample for cortisol measurements and a blood sample to measure several markers of immune function at four different time points: before medical treatment, after medical treatment and before randomization to MBSR or waiting, after the completion of MBSR as well as at 3-month follow-up. A sub-sample will complete a series of tasks while undergoing functional magnetic resonance imaging before and after participation in MBSR.

The primary outcome is pain interference. The investigators will compare the proportion of participants who report reduced pain-related disability, as measured by the Brief Pain Inventory-Interference Scale, in each group. The primary hypothesis is that at 3-month follow-up, there will be at least 30% more responders (≥1.0 decrease in mean Brief Pain Inventory Interference score) in the interdisciplinary program in comparison to medical treatment alone.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* 18 years or older.
* Completed treatment for breast cancer a minimum of 1 year prior to study enrollment.
* Have been experiencing neuropathic pain following their cancer treatment for a minimum of 6 months.
* Report pain intensity levels ≥4 (moderate to severe).

Exclusion Criteria:

* Metastatic disease or current evidence of cancer recurrence
* Pregnancy or breastfeeding
* Unable to complete questionnaires in English or French.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-10; Primary Completion 2017-10 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain-related disability, as measured by the Brief Pain Inventory - Pain Interference scale, at 3-month post-intervention. | Baseline and 3 months post-intervention
  The primary outcome is pain-related disability, as measured by the Brief Pain Inventory - Pain Interference scale. The Brief Pain Inventory (BPI) - Pain Interference consists of 7 numerical scales (0 to 10) rating pain interference with general activity, mood, walking ability, work, relations with other people, sleep and enjoyment of life.

SECONDARY OUTCOMES:
Change from baseline in neuropathic pain intensity, as measured by the Neuropathic Pain Symptom Inventory, at 3 months post-intervention | Baseline and 3 months post-intervention
  Neuropathic pain intensity will be measured using the Neuropathic Pain Symptom Inventory (NPSI), a self-report questionnaire that consists of 10 pain descriptors and two temporal items. Responses are rated on a numerical scale (0-10) and a total intensity score is calculated. Five sub-scores are also derived: spontaneous burning pain, spontaneous pressing pain, paroxysmal pain, evoked pain and paresthesia/dysesthesia.
Change from baseline in pain severity, as measured by the Brief Pain Inventory - Pain Severity scale, at 3 months post-intervention | Baseline and 3 months post-intervention
  Pain Severity will be measured using the Brief Pain Inventory (BPI) - Pain Severity. The BPI consists of 4 numerical scales (0 to 10) rating pain severity at its worst, at its least, on average, and at the time of filling out the measure. Each severity question is analyzed individually.
Change from baseline in mood states, as measured by the Profile of Mood States scale, at 3 months post-intervention | Baseline and 3 months post-intervention
  The Profile of Mood States (POMS-2A) will be used to measure mood disturbance. Participants are asked to rate 65 adjectives using a 5-point likert scale ( 0= not at all, to 4 = extremely) based on how they have been feeling during the past week, including the day they are filling out the questionnaire. A total mood disturbance score is calculated, as well as scores for 6 subscales: depression, tension-anxiety, anger-hostility, vigor-activity, fatigue, confusion-bewilderment.
Overall change in status from baseline, as measured by Patient Global Impression of Change scale, at 3 months post-intervention | Baseline and 3 months post-intervention
  The participants' perceived degree of change in overall status will be measured using the Patient Global Impression of Change (PGIC) scale. The PGIC uses a 7-point likert scale (very much worse, to very much better) to measure how much the participant feels their overall status has changed since the start of the study.
Change from baseline in stress, as measured by the Perceived Stress Scale, at 3 months post-intervention | Baseline and 3 months post-intervention
  The Perceived Stress Scale (PSS) will be used to measure the participants' perceived stress levels. The PSS uses a 5-point likert scale (0=Never, to 4=Very often) to measure the degree of stress a participant has experienced over the past month. A total perceived stress score is obtained by reversing the scores on items 4, 5, 7, and 8, and then summing across all 10 items. Higher scores indicate higher perceived stress.
Change from baseline in depressive symptoms, as measured by the Patient Health Questionnaire - 9 scale, at 3 months post-intervention | Baseline and 3 months post-intervention
  The Patient Health Questionnaire - 9 (PHQ-9) is a 9-item scale used to assess the severity of depressive symptoms over the past two weeks and is based on Diagnostic and Statistical Manual (DSM-IV) diagnostic criteria for major depression. Total scores range from 0 to 27, and clinical cut-points correspond to mild, moderate, moderately severe, and severe depression.
Change from baseline in pain catastrophizing, as measured by the Pain Catastrophizing Scale, at 3 months post-intervention. | Baseline and 3 months post-intervention
  The Pain Catastrophizing Scale (PCS) is a 13-item instrument which will evaluate the degree to which patients have negative self-statements and catastrophizing thoughts and ideations when in pain. The PCS uses a 5-point likert scale (0=not at all, 4=all the time) and consists of three subscales (rumination, magnification, helplessness).
Change from baseline in mindfulness, as measured by the Five Facet Mindfulness Questionnaire, at 3 months post-intervention. | Baseline and 3 months post-intervention
  Mindfulness will be measured using the Five Facet Mindfulness Questionnaire (FFMQ). The FFMQ is a 39-item instrument measuring five aspects of mindfulness: Non-reactivity to inner experience, observing, describing, acting with awareness, and non-judging of experience. Participants are asked to use a 5-point Likert-type scale (1 = never or rarely true; 5 = very often or always true) to rate how true of them they believe each statement to be.
Change from baseline in quality of life, as measured by the Short-Form-12 Health Survey, at 3 months post-intervention. | Baseline and 3 months post-intervention
  Quality of life will be measured by the Short-Form-12 Health Survey (SF-12v.2). The SF-12v2 is a brief, twelve-item self-report measure based on the Short-Form-36. It includes items assessing eight health domains, such as bodily pain, social functioning, role limitations due to physical health, and general health perceptions. Two summary scores, the physical composite scale (PCS) and mental composite scale (MCS) are computed based on the 12 items. Scores range from 0 to 100, with higher scores indicating greater quality of life.
Change from pre-intervention in biomarkers of stress, as measured by hair cortisol levels, at 3 months post-intervention. | Pre-intervention and 3 months post-intervention
  Cortisol is a useful biomarker of stress levels. One cm hair samples will allow us to collect data on cortisol exposure over the past month.
Change from baseline in immune function, as measured by blood levels of interleukin-4, interleukin-6, interleukin-10, tumor necrosis factor - alpha, and C reactive protein, at 3 months post-intervention. | Baseline and 3 months post-intervention
  Six mL whole blood samples will be obtained from participants and the measurement of cytokine secretion and CRP will be performed. The concentrations of interleukin-4 (IL-4), interleukin-6 (IL-6), interleukin-10 (IL-10), tumor necrosis factor - alpha (TNF-α), as well as C reactive protein (CRP) production will be quantified and recorded. All samples and standards will be analyzed in duplicate.
Change from baseline in biomarkers of stress, as measured by telomere length, at 3 months post-intervention. | Baseline and 3 months post-intervention
  Total genomic DNA will be extracted from 0.2 mL of whole blood. The relative average Telomere Length (TL) will be determined and recorded. Samples will be analyzed in triplicate.
Change from pre-intervention in neuronal health, as measured by white matter integrity, at 2 weeks post-intervention. | Pre-intervention and 2 weeks post-intervention
  Changes in participants' neuronal health will be measured with MRI sessions that include diffusion tensor imaging (DTI). These imaging sessions will provide measures of white matter integrity (fractional anisotropy, mean diffusivity, radial diffusivity).
Change from pre-intervention in brain areas associated with emotional regulation, as measured by blood flow in the brain seen in functional magnetic imaging, at 2 weeks post-intervention. | Pre-intervention and 2 weeks post-intervention
  Changes in blood flow to areas of participants' brains known to be associated with emotional regulation will be measured using functional magnetic imaging (fMRI).
Change from pre-intervention in brain structure, as measured by changes in structural volume different areas of the brain, at 2 weeks post-intervention. | Pre-intervention and 2 weeks post-intervention
  High resolution magnetic resonance imaging will be used to look at the anatomy of participants' brains and measure changes in structural volume.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Poulin, PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No